CLINICAL TRIAL: NCT01803217
Title: AV-Hysteresis Versus Mode Switch to AAI (MVP) for the Avoidance of Unnecessary Right Ventricular Pacing
Brief Title: Evaluation of Pacemaker Algorithms to Avoid Unnecessary Right Ventricular Pacing
Acronym: ADVANTAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Klinikum Bamberg (Other); Krankenhaus Peißenberg (Unknown); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GER-EP-010
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Pacemaker Implantation for Sinus Node Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- mode switch to atrial pacing (Experimental)
  Interventions: Other: pacemaker programming to mode switch to atrial pacing versus atrioventricular hysteresis function
- atrioventricular hysteresis function (Active Comparator)
  Interventions: Other: pacemaker programming to mode switch to atrial pacing versus atrioventricular hysteresis function

INTERVENTIONS:
Other: pacemaker programming to mode switch to atrial pacing versus atrioventricular hysteresis function

SUMMARY:
Unnecessary right ventricular pacing has been shown to be detrimental in recipients of implantable pacemaker or defibrillators.

The ADVANTAGE study evaluates the efficacy of two pacemaker based algorithms (atrioventricular hysteresis function versus mode switch to atrial pacing) to reduce right ventricular pacing.

DETAILED DESCRIPTION:
Comparison of the effect of an atrioventricular hysteresis function with a mode switch to atrial pacing on the right ventricular pacing percentage in a multi-centre, prospective, randomized, single blinded, cross-over study.

ELIGIBILITY:
Inclusion Criteria:

Indication for the implantation of a dual-chamber pacemaker

Exclusion Criteria:

Persistent or permanent atrial tachyarrhythmias atrioventricular block 2nd or 3rd degree indication or the implantation of an defibrillator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Right ventricular pacing percentage | 3 months

SECONDARY OUTCOMES:
BNP levels | 3 months

OTHER OUTCOMES:
Occurrence of atrial tachyarrhythmias | 3 months

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Klinikum Bamberg, Bamberg, Bavaria
  - Deutsches Herzzentrum München, Klinik für Herz- und Kreislauferkrankungen, München, Bavaria
  - Krankenhaus Peißenberg, Peißenberg, Bavaria